CLINICAL TRIAL: NCT06818058
Title: A Phase II Multicentric, Randomized, Double-blind, Placebo-controlled Study of TAR-0520 Gel in EGFR Inhibitor-induced Folliculitis.
Brief Title: TAR-0520 Gel in EGFR Inhibitor-induced Folliculitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tarian Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TARIAN 007; 2024-516339-28-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-23; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: EGFR Inhibitor-associated Rash
Keywords: EGFR inhibitor-induced skin rash;; EGFR inhibitor-induced folliculitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active arm (Experimental): Brimonidine tartrate gel
  Interventions: Drug: Brimonidine tartrate Gel
- Placebo arm (Placebo Comparator)
  Interventions: Drug: Placebo gel (no Brimonidine tartrate)

INTERVENTIONS:
Drug: Brimonidine tartrate Gel — Once daily applications for 7 days
  Arms: Active arm
Drug: Placebo gel (no Brimonidine tartrate) — Once daily applications for 7 days
  Arms: Placebo arm

SUMMARY:
A Phase II, multicentric, randomized, double-blind, placebo-controlled, parallel- group trial to confirm the good safaty profile and to explore the preventive effect of topically applied TAR-0520 gel on folliculitis developed in metastatic colorectal cancer (mCRC) patients treated with monoclonal anti-EGFR antibodies.

DETAILED DESCRIPTION:
Cetuximab and panitumumab hae become the standard treatment for patients with metastatic colorectal cancer without RAS gene mutation. Hoever, these EGFR inhbitors induce a broad spectrum of cutaneous toxicities (skin side effects) in 75-90% of patients, including the folliculitis involving the face,upper torso and scalp. The folliculitis appears within 1-2 weeks of anti-EGFR therapy and peaks around 3-5 weeks of treatment. There is no approved treatment to prevent or treat EGFR-induced folliculitis. Tarian Pharma has developed a new topical treatment of EGFRi-induced folliculitis.This study aims to confirm the good safety of TAR-0520 gel in colorectal cancer patients treated with cetuximab or panitmumab and eplore , in the same patients , the effect of TAR-0520 gel on the extent and severity of EGFRi-induced folliculitis.

Patients aged 18 years and over with metastatic colorectal carcinoma planned to be treated with cetuximab or panitumumab injections will be included in the study.

Participants will be randomly allocated to receive either the topical active TAR-0520 gel or its vehicle.The study will include a 7days treatment period with once daily applications of the test product followed by a treatment free period until the start of the next chemotherapy cycle usually 7 days later.The study will cover 4 complete chemotherapy cycles, thus lasting at least 56 days.

ELIGIBILITY:
Inclusion Criteria:

* male or female, who is at least 18 years of age or older at the screening visit
* patients with clinical diagnosis of metastatic colorectal carcinoma planned to be treated with cetuximab or panitumumab injections as part of the chemotherapy protocol
* patients who can understand and sign the Informed Consent Form, can communicate with investigator,can understand and comply with requierements of the protocol, and can apply the study gel by himself/herself or have giver who can apply the product
* patients with predicted life expectency of > 3 months
* patients willing and able to comply with all of the time commitements and procedural requirements of the clinical trial protocol

Exclusion Criteria:

* patients with medical history of EGFR treatment in the past 2 years
* patients with any underlying physical ,psychological or medical condition that, in the opinion of the invstigator, would make it unlikely that the patient will comply with the protocol or complete the study protocol
* patients with any uncotrolled or serious disease, or any medical or surgical condition,that may put the subject at significant risk (according to the investigator's judgement) if he/she participates in the clinical trial
* patients with history of other skin disorders (eg.atopic dermatitis,psoriasis,recurrent skin infections), or a history of illness that, in the opinion of the investigator, would confound the results of the study
* patients with significant skin disease other than EGFRi-induced folliculits within the same body areas planned for study drug application
* patients with a beard that would interfere with administration of the study drug and assessement of study endpoints
* patients with active infection within the treatment area ot in other body areas that requieres initiation of systemic antibiotics
* patients with known or suspected allergies or sensitivities to any components of the study drugs
* female patients who are pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of Treatment - emergent Advers Events (TEAEs) | At Baseline and then at Day 14, Day 28, Day 42 and Day 56 .
  TEAEs will be tabulated in frequency tables by System Organ Class and Preferred Term, based on the Medical Dictionary for Regulatory Activities (MedDRA). Additional summary tables will be provided for AEs that are considered serious (SAEs), related to the study drug, adverse events of special interest (AESIs), and AEs leading to discontinuation.
  The safety conclusions will be based on the comparative analysis of the AEs reported in the two treatment arms.

SECONDARY OUTCOMES:
Efficacy of TAR-0520 gel to prevent EGFR-induced folliculits | The measurements will be performed at Baseline visit and then at Day 14,Day 28,Day 42 and Day 56.
  The preventive effectivness of TAR-0520 gel will be measured by assessing EGFR-induced folliculitis severity using a modified Common Terminology Criteria for Adverse Events (CTCAE) scale (Grade 0-no folliculitis - Grade 4-severe folliculitis)

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hopital Privé Jean Mermoz, Lyon
  - Institut Paoli Calmette, Marseille
  - Centre Antoine Lacassagne, Nice

IPD SHARING:
Plan to Share IPD: No